CLINICAL TRIAL: NCT02472470
Title: Efficacy and Biological Targets of Response to rTMS Therapy in Youth Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Faranak Farzan, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: # 076/2014-01
Record Dates: First submitted 2015-06-10; First posted 2015-06-15 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Depressive Symptoms
Keywords: rTMS; Depression; Youth; TBS; Brain Stimulation; Electrophysiology; Imaging
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): intermitten TBS (iTBS) rTMS applied to the left Dorsolateral Prefrontal Cortex (DLPFC) + continuous TBS (cTBS) rTMS applied to the right DLPFC. The order will be counterbalanced. Administration of this treatment takes roughly 10 minutes. This treatment will be applied daily, 5 days/week, for 2 weeks.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Participants will receive 10 active TBS rTMS sessions once daily on weekdays for 2 weeks.
  Other Names: TBS

SUMMARY:
Youth depression is a debilitating disorder that exacts enormous social, economic and personal cost. Unfortunately, treatments which are conventionally used to treat adult depression have often modest to no efficacy in youth and have side effects. Thus, there is a tremendous imperative to develop new treatments for youth depression. Investigators propose to examine the efficacy of a short form of repetitive transcranial magnetic stimulation (rTMS) for youth depression and examine its biological targets. This will be the first study examining the efficacy of a short rTMS protocol in youth diagnosed with depression who fail responding to or are intolerable to antidepressants. If the results are positive, investigators will have identified a novel treatment that may be both more efficacious, better tolerated and more acceptable treatment for youth depression. Finally, identifying the biological mechanisms leading to treatment efficacy will lead to more personalized treatments for youth depression and will be groundbreaking vis à vis understanding the mechanisms involved in this illness.

DETAILED DESCRIPTION:
The highest rates of depression are reported in youth 16-24 years of age and youth depression is a significant source of burden to the individual, their families, and to society. Unfortunately, current treatments (e.g., selective serotonin reuptake inhibitors), which are conventionally used to treat depression often have modest and sometimes no efficacy in youth. Also, accumulating evidence suggests that these medications may increase suicidal thoughts in adolescents and young adults below the age of 24. In addition to pharmacological treatments, cognitive behavioral therapy (CBT) has been used alone or in combination with medications for treating depression in this age group. Although randomized controlled trials and practice guidelines support the use of CBT alone and CBT with an antidepressant medication for adolescent depression, a large minority of adolescents do not respond to either treatment approaches.Thus, there is a tremendous imperative to develop new treatments for youth depression.

Investigators propose to examine the efficacy of repetitive transcranial magnetic stimulation (rTMS) for youth depression. There are several reasons for pursuing this treatment: 1) rTMS applied to the dorsolateral prefrontal cortex (DLPFC), a cortical region implicated in pathophysiology of depression, is a safe and FDA approved treatment for adults with medication-resistant depression; 2) Young age is suggested to be a good predictor of response to rTMS treatment; 3) rTMS trials in adolescence and youth with medication resistant depression provide evidence that rTMS is a safe efficacious and well tolerated treatment for adolescents that does not increase suicidal thoughts. Additionally, recently rTMS parameter developments such as theta burst stimulation (i.e., TBS) provide compelling evidence for efficacy in less of the time it takes to administer conventional rTMS, thus lowering the overall costs and increasing the number of patients that can be treated.

It is imperative that research investigate treatment related biological mechanisms, such that increases in understanding can lead to enhanced efficacy. Investigators will utilize a novel and powerful in vivo brain mapping technique of TMS combined with electroencephalography (TMS-EEG) that permits non-invasive assessment of inhibitory, connectivity and plasticity mechanisms from the DLPFC. The pathophysiology of depression has been linked to impairment in neural plasticity and connectivity and neural and behavioral inhibition - mechanisms that can be measured through TMS-EEG and maybe changed by TBS treatment. Therefore, investigating the association between TBS-related changes in plasticity, connectivity and inhibition may be key to understanding both the treatment mechanisms involved in youth depression and predictors of treatment response in this disorder.

Therefore the specific aims in this study are twofold:

1. To examine the efficacy of TBS applied to the DLPFC for youth depression, and
2. To identify biological targets and predictors of response to TBS applied to the DLPFC for youth depression.

ELIGIBILITY:
Inclusion Criteria:

* outpatients
* between the ages of 16 and 24
* competent to consent to study participation
* Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of MDD single or recurrent
* no change in treatment (psychotherapy or medication) for at least four weeks prior to participation in the study
* HRSD-17 score of 20 and higher
* at least one failed/refused/intolerant to antidepressant trial in the current episode as determined by Antidepressant Treatment History Form (ATHF)
* No safety concerns endorsed on TMS Screening and Information Form

Exclusion Criteria:

* lifetime MINI diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, delusional disorder, current psychotic symptoms, post traumatic stress disorder, obsessive compulsive disorder, autism spectrum disorder, a history of epilepsy or any other major neurological disorder
* history of substance use disorders (moderate to severe) within the last 3 months as determined by MINI
* concomitant major unstable medical illness
* acutely suicidal or high risk for suicide as assessed by a study psychiatrist
* not eligible to receive TMS or MRI as indicated by TMS Screening and Information Form
* a change in treatment status during the study trial that will be considered a confound to the study. This includes change in medication or Cognitive Behavioral Therapy, each reviewed case by case by the study psychiatrists.
* medications that are considered a confound to the study including benzodiazepines, antipsychotics, mood stabilizers, stimulants and anticonvulsants.
* missing more than 20% of the treatment sessions consecutively (i.e., 2 sessions in a row) or 40% (i.e., 4 sessions) within two weeks
* have failed brain stimulation in the past

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms as Measured by HRSD-17 | Baseline (before treatment trial starts), week 1 (after 5 days of treatment), and week 3 (within a week after the end of the 2-week treatment trial)
  Outcome measure is measured by a change in the HRSD-17 score from baseline to week 1 and week 3. A 50% improvement in the score is considered response to rTMS

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | Baseline (before treatment trial starts), week 1 (after 5 days of treatment), and week 3 (within a week after the end of the 2-week treatment trial)
Children's Depression Rating Scale, revised-version (CDRS-R) | Baseline (before treatment trial starts), week 1 (after 5 days of treatment), and week 3 (within a week after the end of the 2-week treatment trial)
  Only in participants under 18 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Faranak Farzan, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dhami P, Moreno S, Croarkin PE, Blumberger DM, Daskalakis ZJ, Farzan F. Baseline markers of cortical excitation and inhibition predict response to theta burst stimulation treatment for youth depression. Sci Rep. 2023 Nov 4;13(1):19115. doi: 10.1038/s41598-023-45107-1. PMID 37925557
- [Derived] Dhami P, Atluri S, Lee J, Knyahnytska Y, Croarkin PE, Blumberger DM, Daskalakis ZJ, Farzan F. Neurophysiological markers of response to theta burst stimulation in youth depression. Depress Anxiety. 2021 Feb;38(2):172-184. doi: 10.1002/da.23100. Epub 2020 Oct 1. PMID 33001549
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research